CLINICAL TRIAL: NCT07120906
Title: Augmented Reality Real-Time Guidance for MRI-Guided Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Woodrum, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-011504
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MR-guided needle placement (Experimental): An augmented reality display compatible with MRI will be used to assist with guidance of needle placement for biopsy or ablation procedure.
  Interventions: Device: MRI guided procedure software evaluation

INTERVENTIONS:
Device: MRI guided procedure software evaluation — For the use of the MRI-needle guidance system (LUMENA) developed by CLEAR GUIDE MEDICAL during clinical MRI-guided needle placement procedures for patients undergoing a liver biopsy/procedure.

SUMMARY:
The purpose of this research is to evaluate the safety and feasibility of using a needle guidance system (LUMENA) create by CLEAR GUIDE MEDICAL for needle placement for biopsy or liver tumor ablation procedures.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the safety and feasibility of using a needle guidance system (LUMENA) create by CLEAR GUIDE MEDICAL for needle placement for biopsy or liver tumor ablation procedures.

The MRI compatible guidance system will not change the needle biopsy or ablation procedure but will provide the doctor doing the procedure with an augmented reality display to better track the needle path as it is being inserted in the target. Otherwise, the procedure will be carried out in the same manner as it is currently done under MRI or CT or X-ray guidance.

Participants who have been scheduled for the guided biopsy or ablation procedure of the liver will be invited to take part in this research.

Study participation involves one study visit. Participants will be in the study until the biopsy or ablation procedure is completed. The biopsy procedure will take approximately 60 minutes to complete. The ablation procedure will take approximately 4 hours to complete.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, ages 18-90 years
* Patient referred to Interventional Radiology for image-guided liver needle placement for ablation/biopsy.

Exclusion Criteria:

* Patients who are unable to give informed consent themselves or through their parents.
* Patients that do not fit into MR scanner (70 cm bore) with room for needle placement.
* Contraindications to MRI such as MR-unsafe implants.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | Baseline (during procedure)
  Use of the guidance system will be considered feasible if the system is used successfully in more than 80% of procedures
Safety of intervention (adverse events) | Up to 4 hours
  Participants will be monitored for adverse events during the procedure and during recovery time following the procedure. The intervention will be considered safe if the needle is successfully placed in the target with no serious adverse events and total adverse events <10%.

SECONDARY OUTCOMES:
Number of needle passes | Baseline (during procedure)
  Recorded during the procedure by a member of the technical staff who will be there monitoring use of the guidance system.
Procedure time | Baseline (during procedure)
  Procedure time will be recorded. Start time will be when initial imaging is obtained (planning image). The end time will be when the final imaging is taken (needle placement completed).
Accuracy of needle placement | Baseline (during procedure)
  Assessed using MRI images showing needle placement, planned versus actual.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Woodrum, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials